CLINICAL TRIAL: NCT04491734
Title: Open Label Tolerability Study of a Novel Microbiome Therapeutic (ISOT-101), Maltosyl-Isomalto-oligosaccharides (MIMO), in Subjects With Gastroesophageal Reflux Disease
Brief Title: Tolerability Study of a Novel Microbiome Therapeutic in Subjects With Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ISOThrive Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1001
Record Dates: First submitted 2020-06-23; First posted 2020-07-29 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Gastroesophageal Reflux
Keywords: GERD; reflux; remote; PPI
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tolerability Arm (Other): Single arm study of active study product
  Interventions: Dietary Supplement: maltosyl-isomalto-oligosaccharides (MIMO)

INTERVENTIONS:
Dietary Supplement: maltosyl-isomalto-oligosaccharides (MIMO) — Digestion-resistant carbohydrate, ISOT-101, a specific formulation of maltosyl-isomalto-oligosaccharides (MIMO), that serves as a prebiotic, feeding selected bacteria that commonly inhabit the human GI tract.

SUMMARY:
This is a remote study. No office visits required. The purpose and efficacy endpoint of this study is to assess whether GERD patients tolerate ISOT-101. In addition, usage of the ReQuest validated questionnaire to measure GERD symptoms will be explored as well as usage of the validated SF-36 quality of life (QoL) questionnaire. Each subject serves as his/her own control. Relative tolerability in subjects both on and off proton pump inhibitors (PPIs) will be compared. Subjects naive to PPIs, currently taking PPIs and historically on PPIs will be evaluated with ReQuest and QoL scores. In addition, survey measurements will be taken on a subset of 10 subjects that are non-responders to PPIs. These will not be included in the statistical analysis with the above groups. A tertiary endpoint of this study is to assess any relevant adverse events that occur.

DETAILED DESCRIPTION:
Introduction and Background GERD is found in about one-third of the population of the USA. About 20 to 45 million people have been diagnosed by a doctor and have been prescribed daily acid reducing medications called proton pump inhibitors (PPIs), which are the mainstay of medical therapy for GERD. PPIs don't cure GERD and many patients take them indefinitely for adequate symptom control. In addition, clinicians and researchers have identified concerns with regard to chronic PPI use and the resulting possible adverse effects due to chronic diminished gastric acid production. The potential adverse effects with reasonable association to PPIs include osteoporosis, fractures, pneumonia, C. difficile colitis, small intestinal bacterial overgrowth (SIBO), hypomagnesemia, vitamin B-12 deficiency, and iron deficiency anemia. The frequent claims of potential PPI adverse effects that appear in public media has also worried patients. In a recent article, 46% of patients on PPIs want to discontinue them and 39% unfortunately have tried to do so without medical advice, increasing the risk of GI bleeding, Barrett's esophagus and esophageal adenocarcinoma. Other patients, such as those at risk for C. difficile infection, osteoporosis (the elderly), patients with small intestinal bacterial overgrowth, among others, should not be on PPIs indefinitely. Unfortunately, there has been no reliable cure or adequate alternative that does not share adverse effects. ISOThrive has produced a proprietary digestion-resistant carbohydrate, ISOT-101, a specific formulation of maltosyl-isomalto-oligosaccharides (MIMO), that serves as a prebiotic, feeding selected bacteria that commonly inhabit the human GI tract. MIMO has an FDA Generally Recognized As Safe (GRAS) status. Since the dawn of agrarian societies, grains were converted to bread using a sourdough fermentation process. MIMO molecules are generally found in such breads. These forms of breads and other sources of MIMO have been inadvertently removed from the daily diet and so can no longer feed selective bacteria that may have played a protective role for prior generations.

Study Rationale This is a remote study. No office visits required. The purpose and efficacy endpoint of this study is to assess whether GERD patients tolerate ISOT-101. In addition, usage of the ReQuest validated questionnaire to measure GERD symptoms will be explored as well as usage of the validated SF-36 quality of life (QoL) questionnaire. Each subject serves as his/her own control. Relative tolerability in subjects both on and off proton pump inhibitors (PPIs) will be compared. Subjects naïve to PPIs, currently taking PPIs and historically on PPIs will be evaluated with ReQuest and QoL scores. In addition, survey measurements will be taken on a subset of 10 subjects that are non-responders to PPIs. These will not be included in the statistical analysis with the above groups. A tertiary endpoint of this study is to assess any relevant adverse events that occur.

Study Design The test material is ISOT-101. It is an approximately 90% pure maltosyl-isomalto-oligosacchride (MIMO) prebiotic syrup produced by bacterial fermentation/bio-conversion of sucrose and maltose. It is taken 1g daily at bedtime.

Subjects will have been previously diagnosed with GERD and will fall into one of the following four groups:

1. Symptomatic subjects currently not taking PPI therapy and who are naive to PPIs.
2. Symptomatic subjects currently not taking PPI therapy who were responsive to prior PPI therapy (either QD or BID) and who have been off PPIs for at least four weeks.
3. Symptomatic subjects currently taking PPI therapy (either QD or BID) who are partial responders to PPIs.
4. 10 symptomatic subjects who have had no benefit from PPIs and have not taken PPIs for at least 4 weeks.

All subjects will have active GERD symptoms as determined by the ReQuest validated GERD specific questionnaire. The study has been designed to have each subject serve as their own control so there will be no placebo arm. Each subject will receive ISOT-101 according to the protocol. Recruitment for subjects with GERD will be by referrals from GI specialists, primary care physicians and general advertising. Each candidate will be given information as to how to contact the study coordinator to enroll in the study. The goal is to assess 110 subjects after the Screening Phase, including the 10 subjects who did not respond to PPIs. All subjects will be screened per the eligibility criteria delineated in this protocol by the study coordinator.

Two phases have been designed into this study. Phase 1 is the Screening Phase (SP). Phase 2 is the Tolerability Phase (TP). Subjects will be instructed to take a daily GERD symptom questionnaire, the ReQuest Short Version, daily throughout the study. At five timepoints, specific scores will be established for comparison and statistical analysis. These timepoints are: (1) SP7 - baseline on current therapy (if any) without ISOT-101; (2) TP7 - 1 week on both current therapy (if any) and ISOT-101; (3) TP14 - 2 weeks on both current therapy (if any) and ISOT-101; (4) TP21 - 3 weeks on both current therapy (if any) and ISOT-101; (5)) TP28 - 4 weeks on both current therapy (if any) and ISOT-101. At each of these timepoints, subjects will also complete the ReQuest Long Version and the SF-36 Health Survey QoL validated questionnaires. They need not complete the ReQuest Short Version on days that the ReQuest Long Version is required. Subjects will report any usage of all GERD medications (PPI, H-2 antagonists, antacid) throughout their study participation.

Enrollment An adequate number of individuals will need to be screened during the Screening Phase, using disease specific validated questionnaires to yield approximately 110 qualified subjects to enter and likely complete the Tolerability Phase of the study. Recruitment may involve primary care physicians and/or gastroenterologists who will make IRB approved study information available to patients who are symptomatic for GERD. Such patients will include those partial responders on PPI therapy; those who responded to PPIs, but have previously stopped their PPI therapy for at least 4 weeks; those who are naive to PPI therapy, and 10 subjects that have had no benefit from PPIs and have not been on PPI therapy for at least 4 weeks. Deviations from the inclusion and exclusion criteria will not be allowed so as not to jeopardize the scientific integrity of the study, regulatory acceptability, or subject safety. Therefore, adherence to the criteria as specified in the protocol is essential.

All subjects will be required to sign an IRB-approved informed consent or e-consent that complies with the requirements of both 21 CRF Part 50 and Health Insurance Portability and Accountability Act (HIPAA) before entering the study.

The duration of the study is defined for each subject as the date a signed written informed consent (or e-consent) is provided through Tolerability Phase Day 28. Total participation in study may last up to 8 weeks. A comparable gender distribution is sought for the final analysis, therefore, the ratio of male to female (or female to male) subjects completing the Tolerability Phase will be capped at 60% of the total.

Concomitant Medications and Washout Periods GERD medications: Subjects currently taking PPI therapy (either QD or BID) who are partial responders to PPIs may continue taking PPIs throughout the study as needed. Subjects not taking PPIs prior to being enrolled may also take PPIs as needed. Antacids or H-2 antagonists may be taken regularly or intermittently as needed throughout the conduct of this study. All GERD-related medications taken by the subject should be recorded daily via the daily electronic survey.

Prebiotic and/or probiotic supplements: Enrolled subjects must stop taking all prebiotic and/or probiotic supplements 2 weeks prior to entering the Screening Phase of the study. Subjects must refrain from taking prebiotic or probiotic supplements through Tolerability Phase Day 28.

Sleep medications: Enrolled subjects taking medications for sleep disorders must be on a stable dose at time of consent and continue at said dose through Tolerability Phase Day 28.

Antibiotics: Subjects must not have taken antibiotics within 6 months prior to signing of consent or at any time during their participation in the study. If antibiotics are prescribed to the subject during study participation, subject must be withdrawn from study and discontinue daily ISOT-101 immediately.

All study product sachets (used and unused) must be returned to Investigator for product accountability.

Subject Study Flow Process

No study-related activities will be performed and no subject data will be collected prior to completion of the informed consent process.

Screening Phase (SP):

To enter the SP, subjects must have previously been diagnosed with GERD, be symptomatic on their current therapy or lack of therapy, and fall into one of the 4 study groups noted in Section 4.0 above. The SP will last for 7 days. Subjects who do not qualify at any point during the SP will not be allowed to move into the Tolerability Phase (TP). The TP will last 28 days, beginning with first dose of ISOT-101.

Following Day 7 of SP, the average of the daily ReQuest Short Version scores will be used to establish a baseline score to confirm that the subject is experiencing GERD symptoms. Any subject who has a ReQuest Short Version (RQ) average score of >= 3.37 (90 percentile) or ReQuest GI (RQ-GI) average score >=0.95 on the will be eligible to transition to the Tolerability Phase. The ReQuest Short Version SP1-SP7 average and SF-36 will serve as a baseline. Investigator will verify eligibility prior to study staff contacting subject.

Once eligibility has been verified by the PI, the study coordinator will inform subject and confirm that subject wishes to continue in the study. Once confirmed, study coordinator will:

* Review concomitant medications
* Collect any adverse events
* Review calendar for remainder of study
* Provide instructions for daily dosing of ISOT-101
* Confirm mailing address
* Arrange for shipment of 30-day supply of ISOT-101 to the subject There may be up to 7 calendar days between SP Day 7 and TP Day 1 depending on length of time to ship/receive ISOT-101.

Tolerability Phase (TP)

Subjects will take their current GERD therapy as follows:

* If on PPI therapy QD or BID, then the PPI is to be taken as the subject customarily has taken it, prior to beginning the study.
* If on an H-2 antagonist or antacid, then the subject may continue these medications as needed throughout the study.

All GERD medications and other medications will be recorded daily via the electronic survey.

• ISOT-101 will be taken daily at bedtime (one sachet per day). This will be the last thing swallowed prior to bedtime (no rinsing, and after brushing teeth) As the primary endpoint, tolerability of ISOT-101 will be assessed. In addition, changes in the ReQuest Short Version GERD symptom scores (RQ, RQ-GI and RQ-WSO) and SF-36 scores will be assessed for all subjects as well as for the sub-group of subjects that completed all 4 weeks of the protocol. Changes in ReQuest symptom scores, or SF-36 scores, between time point 1 and time point 2 will be the basis of this assessment. Further evaluation will include comparison of ISOT-101 tolerability in the 4 subject sub-groups using these two time points.

The safety endpoint of the study is to ensure that any adverse events that are reported or observed during the study are appropriately recorded.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking male and female adults between the ages of 25 and 75, inclusive
2. Body mass index (BMI) <35 and >19
3. Either 3.a. or 3.b. or both, based on the Screening Phase ReQuest Short and Long Version responses:

   1. At least one incidence of (a) acid complaints; (b) upper abdominal/stomach complaints and RQ Total score >3.37 or RQ-GI score >0.95
   2. Four days or more of combined incidence of (a) acid complaints; (b) upper abdominal/stomach complaints.
4. History (minimum of three months) of GERD symptoms as defined in #3 above
5. Must be on stable doses of medications, if any, prescribed for chronic conditions other than GERD
6. If female, must be on an active contraceptive measure or have male partner(s) with suitable protective measures
7. Have access to a computer/tablet/phone with internet access and active e-mail account in order to complete electronic surveys daily throughout study participation
8. Ability and willingness to give consent to participate in study

Exclusion Criteria:

1. Significant comorbidities that are not medically stable
2. History of scleroderma, diabetes, Barrett's esophagus, esophageal cancer, esophageal stricture, or esophageal scarring (fibrosis)
3. Known hiatal hernia > 2cm
4. Positive diagnosis for Helicobacter pylori (HP) or has had an HP infection within 45 days of study entry
5. History of surgery or endoscopic treatment including fundoplication and dilation for esophageal stricture
6. History of gastric surgery (except for endoscopic removal of benign polyps) or bariatric surgery
7. BMI >=35, BMI <=19
8. History of diseases that have symptoms that may be confused with GERD, such as eosinophilic esophagitis, angina, gastritis, esophageal spasm, rumination, or other conditions involving the mouth, throat, chest or abdomen
9. Active history of nicotine use, cannabis use or alcohol abuse (as defined by: greater than 14 drinks/week or 4 drinks/day for men, 7 drinks/week or 3 drinks/day for women). Has used any tobacco, nicotine or cannabis products in the last 6 months or has abused alcohol in the last 6 months
10. Taking any excluded medications listed in the protocol (e.g. metformin, antibiotics within the prior 6 months.)
11. If female, is pregnant, lactating, or intending to become pregnant before, during or within 4 weeks after participating in this study or intending to donate ova during such time period
12. Primary sleep disorder including sleep apnea, restless leg syndrome, or insomnia
13. Colon prep within 30 days prior to study entry
14. Use of any investigational product within 90 days prior to study entry
15. Participation in another investigation (clinical trial) during the course of this study
16. Participation in a rigorous weight loss program or have any planned changes in diet or lifestyle, such as getting married, change in residence, change in job, or other highly stressful event
17. Diagnosis of inflammatory bowel disease, irritable bowel syndrome, or chronic diarrhea (mild chronic constipation is allowed)
18. Employment (or relative of an employee) or involvement in any way with ISOThrive Inc.
19. An investigator, key study personnel or first degree relative of anyone involved with the study
20. Other conditions or situations that, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Tolerability of ISOT-101 using GERD ReQuest Short Version | 4 weeks
  Assess whether symptomatic GERD patients tolerate ISOT-101 by measuring the differences in baseline and post-intervention score using GERD ReQuest Short Version. The scores for weeks 1, 2, 3, and 4 will be compared with baseline. With regard to the ReQuest Short Version questionnaire, the range is 0 to 46.28 with higher numbers reflecting more severe symptoms. Tolerability is defined as the post-intervention score is equal to or less than baseline.
Tolerability of ISOT-101 using GERD ReQuest Long Version | 4 weeks
  Assess whether symptomatic GERD patients tolerate ISOT-101 by measuring the differences in baseline and post-intervention scores using GERD ReQuest Long Version. The scores for weeks 1, 2, 3, and 4 will be compared with baseline. With regard to the ReQuest Long Version, the range is 0 to 46.28 with higher numbers reflecting more severe symptoms. Tolerability is defined as the post-intervention score is equal to or less than baseline.
Tolerability of ISOT-101 using Rand Short Form-36 (v1.0) | 4 weeks
  Assess whether symptomatic GERD patients tolerate ISOT-101 by measuring the differences in baseline and post-intervention scores using Rand Short Form-36 (v1.0). The scores for weeks 1, 2, 3, and 4 will be compared with baseline. The range of the SF-36 scoring is 0-100 with higher numbers defining a more favorable health state. Tolerability is defined as the post-intervention score is equal to or greater than baseline.

SECONDARY OUTCOMES:
Measure adverse events | 4 weeks
  Assess any relevant adverse events

CONTACTS AND LOCATIONS:
Overall Officials: John Selling, MD, Principal Investigator — ISOThrive Inc.
Locations (1):
- ISOThrive Inc., Manassas, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
This study will be conducted in accordance with the International Council for Harmonisation (ICH) E6 R2. The Investigator agrees to maintain adequate documentation for the subjects participating in this clinical research project. The Investigator agrees to maintain accurate case report forms and source documentation as part of the case histories. Subjects will enter their data into the data capture system (REDCap). The analysis data sets will be generated from data captured in REDCap.
  All documents and data shall be produced and maintained in such a way as to assure control of documents and data to protect the subject's privacy as far as reasonably practicable. All attempts will be made to preserve subject confidentiality.